CLINICAL TRIAL: NCT00801970
Title: Fear of Childbirth (Tokophobia) - Etiology, Essence and Clinical Implications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Miki Bloch, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-08-MB-0064-CTIL
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Phobias
Keywords: Fear of childbirth; Tokophobia; Anxiety; Labor; Pregnancy; Cognitive-behavioral; Psychoanalysis; Group Therapy; etiology
MeSH Terms: conditions — Phobic Disorders; Anxiety Disorders | interventions — Psychotherapy; Cognitive Behavioral Therapy; Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 - Pregnant - Tokophobic (Experimental): Psychoanalysis treatment.
  Interventions: Behavioral: Psychological Treatment
- 2 - Pregnant - Tokophobic (Experimental): Cognitive-Behavioral treatment.
  Interventions: Behavioral: Psychological Treatment
- 3 - Non-pregnant - Tokophobic (Experimental): Group Therapy
  Interventions: Behavioral: Group Therapy
- 4 - Control (No Intervention): Pregnant and non-pregnant non-tokophobic women will answer questionnaires. Won't receive therapy.

INTERVENTIONS:
Behavioral: Psychological Treatment — 15 weekly therapy sessions.
  Other Names: Psychotherapy; Psychodynamic therapy; Cognitive Behavioral Therapy; CBT
  Arms: 1 - Pregnant - Tokophobic; 2 - Pregnant - Tokophobic
Behavioral: Group Therapy — 3 months of weekly group therapy sessions.
  Other Names: Psychotherapy; Group Psychotherapy
  Arms: 3 - Non-pregnant - Tokophobic

SUMMARY:
The purpose of this study is twofold:

* to understand the etiology and the essence of fear of childbirth
* to examine the implications and efficiency of several forms of psychological therapy.

DETAILED DESCRIPTION:
Fear of childbirth (Tokophobia) is inconsistently defined in the research literature: some define it as an anxiety disorder while it is often defined as a form of phobia; some regard only the pre-pregnancy period, some regard the anxiety during pregnancy and some focus on the labor process. Despite the high prevalence (between 13%-20% of fertile women), research in this area is scarce and the current findings are incohesive due to various conceptualizations of the phenomenon and to various measurement methods.

ELIGIBILITY:
Inclusion Criteria:

* subjective diagnosis of tokophobia

Exclusion Criteria:

* currently undergoing psychological therapy
* Major Depression
* Acute Anxiety
* Psychosis
* Bipolar Disorder
* Suicidal
* Substance abuse
* Non-compliant personality disorder
* Health problems during pregnancy that affect perception

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-06 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Tokophobia existing and new measures (e.g. Pregnancy anxiety scale, Levin, 1991; Tokophobia subjective scale) | Pre-treatment, Mid treatment, End of treatment

SECONDARY OUTCOMES:
For pregnant subjects - labor preference, duration and pain medication assessment. | post-labor

CONTACTS AND LOCATIONS:
Overall Officials: Miki Bloch, M.D, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Psychiatry Outpatient Clinic - Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Areskog B, Uddenberg N, Kjessler B. Fear of childbirth in late pregnancy. Gynecol Obstet Invest. 1981;12(5):262-6. doi: 10.1159/000299611. PMID 7262639
- [Background] Eriksson C, Jansson L, Hamberg K. Women's experiences of intense fear related to childbirth investigated in a Swedish qualitative study. Midwifery. 2006 Sep;22(3):240-8. doi: 10.1016/j.midw.2005.10.002. Epub 2006 Apr 17. PMID 16603282
- [Background] Hofberg K, Brockington I. Tokophobia: an unreasoning dread of childbirth. A series of 26 cases. Br J Psychiatry. 2000 Jan;176:83-5. doi: 10.1192/bjp.176.1.83. PMID 10789333
- [Background] Hofberg K, Ward MR. Fear of childbirth, tocophobia, and mental health in mothers: the obstetric-psychiatric interface. Clin Obstet Gynecol. 2004 Sep;47(3):527-34. doi: 10.1097/01.grf.0000132527.62504.ca. No abstract available. PMID 15326415
- [Background] Alehagen S, Wijma K, Wijma B. Fear during labor. Acta Obstet Gynecol Scand. 2001 Apr;80(4):315-20. doi: 10.1034/j.1600-0412.2001.080004315.x. PMID 11264605
- [Background] Eriksson C, Westman G, Hamberg K. Experiential factors associated with childbirth-related fear in Swedish women and men: a population based study. J Psychosom Obstet Gynaecol. 2005 Mar;26(1):63-72. doi: 10.1080/01674820400023275. PMID 15962723
- [Background] Johnson R, Slade P. Does fear of childbirth during pregnancy predict emergency caesarean section? BJOG. 2002 Nov;109(11):1213-21. doi: 10.1046/j.1471-0528.2002.01351.x. PMID 12452457
- [Background] Olde E, van der Hart O, Kleber R, van Son M. Posttraumatic stress following childbirth: a review. Clin Psychol Rev. 2006 Jan;26(1):1-16. doi: 10.1016/j.cpr.2005.07.002. Epub 2005 Sep 19. PMID 16176853
- [Background] Saisto T, Halmesmaki E. Fear of childbirth: a neglected dilemma. Acta Obstet Gynecol Scand. 2003 Mar;82(3):201-8. PMID 12694113